CLINICAL TRIAL: NCT02786589
Title: Clinical Study of Plasmodium Immunotherapy for Advanced Non-small Cell Lung Cancer
Brief Title: Plasmodium Immunotherapy for Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Collaborators: CAS Lamvac Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ming Ou-Yang, Associate Chief Physician, State Key Laboratory of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KLRD-L-001
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: Lung cancer Immunotherapy; Plasmodium vivax; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood-stage infection of P. vivax (Experimental): This is a single arm study that enrolls 30 patients to receive Plasmodium immunotherapy.
  Interventions: Biological: Blood-stage infection of P. vivax

INTERVENTIONS:
Biological: Blood-stage infection of P. vivax — Each patient will be vaccinated with P. vivax-infected red blood cells containing approximately 0.3-1×10^7 Plasmodium parasites.And successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples.The treatment will last at least 12 weeks from the day of finding the Plasmodium from peripheral blood and will be terminated by chloroquine phosphate or Artemisinin compound preparation or Artesunate injection.

SUMMARY:
The objective of this study is to evaluate the safety and the effectiveness of Plasmodium immunotherapy (blood-stage infection of Plasmodium vivax) for advanced non-small cell lung cancer.The treatment will last 3-6 months from the day of successful infection and will be terminated by antimalarial drugs.

DETAILED DESCRIPTION:
In our study，30 patients with stage III/IV NSCLC will be enrolled to receive vaccination with an optimal concentration and amount of blood-stage P. vivax to observe the infection time, rate and cycle; principal clinical symptoms such as fever and anemia; heart, liver and kidney function; changes in spleen morphology and function, and dynamic changes in the function of peripheral immune cells. Moreover, the patient's tolerance to Plasmodium infection and changes in tumor-related parameters will be observed.

The duration of the planned treatment is 3-6 months, and successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples. The treatment will last at least 12 weeks from the day of finding the Plasmodium from peripheral blood and will be terminated by chloroquine phosphate or Artemisinin compound preparation or Artesunate injection. Each patient will be vaccinated with P. vivax-infected red blood cells containing approximately 0.3-1×10^7 Plasmodium parasites. After vaccination, the onset and duration of peripheral parasitemia and the infection rate; principal clinical symptoms such as Chills, fever, pain (headache, joint pain, etc.), digestive tract reaction;peripheral hemogram changes；heart, liver and kidney function; changes in lung function, and dynamic changes in the function of peripheral immune cells will be observed. Moreover, the patient's tolerance to Plasmodium infection and changes in tumor-related parameters will be observed.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age, male or female
* Unresectable stage III or IV non-small cell lung cancer, diagnosed by histological and radiological findings (UICC, Seventh Ed.), and of any histological subtype. Cancer staging during the initial diagnosis must be confirmed by radiographic findings (CT and/or MRI and/or PET-CT)
* During study treatment, the patient should not receive other treatments, including chemotherapy, radiotherapy, targeted therapy, other biological therapy, physical therapy, traditional Chinese medicine, and so on
* At least 5 half-life of the targeted drug (the half- life calculation is based on the targeted drug instructions) since the end the targeted therapy;More than 12 weeks since the end of radiotherapy or chemotherapy (common or continuous)
* Expected survival > 16 weeks
* ECGO score of 0 or 1
* PLT ≥100 × 10^9/L, WBC ≥ 4 × 10^9/L, and HGB ≥ 100 g/L; no significant morphological abnormalities of red blood cells, or anemia (iron deficiency anemia, autoimmune hemolytic anemia, thalassemia, etc.)
* The patient's peripheral blood immune cell count and immune function test are close to normal or normal, and the heart and lungs and kidneys are normal.
* The patient is willing to receive Plasmodium immunotherapy and is able to sign the informed consent
* For female patients: the result of a pregnancy test must be negative at screening. All subjects must consent to use birth control methods during treatment and for two months after discharge
* The subject is willing to follow the in-hospital exam and treatment and follow-up schedule
* The patient can return for regular scheduled follow-up visits during the 2-year follow-up period
* The subject agrees that the investigators may report and publish the results of this clinical study

Exclusion Criteria:

* Total ≤ 4 weeks after surgical treatment or other forms of treatments
* Active chronic lung diseases (hypoxemia due to bronchial asthma, tuberculosis, other conditions); lung metastatic tumor; other comorbid tumors
* Patients with newly diagnosed brain metastasis (not including the previous brain metastatic lesion, which is not visible by image at the time of screening)
* Patients with autoimmune disease or other immunodeficiency diseases
* Patients taking long-term steroids or immunosuppressants
* Patients with severe hemoglobin disease or severe G6PD deficiency
* Patients with active or chronic symptomatic hepatitis
* Patients with other serious complications such as severe hemoptysis and massive pleural and ascitic fluid
* Liver impairment: ALT > 2.5 x ULN, AST > 2.5 x ULN, bilirubin > 1.5 x ULN
* Renal impairment: serum creatinine ≥ 1.5 x ULN
* Patients with chronic heart disease, primarily those with recent (within a year) myocardial infarction, serious arrhythmias, heart failure, or aortic aneurysm
* Patients with serious drug allergy
* Patients with splenectomy or splenomegaly
* Pregnant and nursing women
* Patients who participating in other clinical trials at the same time or less than 12 weeks since withdraw from other clinical trials
* Any condition that makes the subject ineligible to participate (in the opinion of the investigator)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-27 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v4.0 | 2 years
  Adverse events will be evaluated according to NCI CTCAE 4.0, and the incidence of adverse events will be calculated.

SECONDARY OUTCOMES:
Progression free survival(PFS) | 2 years
  Progression free survival(PFS):Starting from treatment until the disease is first found or the time of any cause of death(disease progression refers to tumor growth, or metastasis of primary tumor, or discovery of new lesions).
Overall survival(OS) | 2 years
  The time starting from the treatment to death of whatever causes (when subjects have lost to follow-up before death , the last follow-up time will be calculated as the time of death).
Tumor marker level | 2 years
  The patient's sensitive tumor markers will be reviewed periodically from the time they are enrolled into the study.
Objective response rate(ORR) | 2 years
  The proportion of patients whose tumor is reduced to a certain amount and maintain a certain period of time.
Quality of life score | 2 years
  Patients are regularly with QLQ-C30(cancer patient quality of life scale)to assess the quality of life of the patients.
Time to progression(TTP) | 2 years
  The time starting from the research to tumor progression.
1 year of survival rate | 2 years
  The number of cancer cases remaining after 1 year of treatment/the total number of cancer cases treated*100%.
2 year of survival rate | 2 years
  The number of cancer cases remaining after 2 year of treatment/the total number of cancer cases treated*100%.
Immunological index | 2 years
  Detection of absolute number of immune cells(such as CD3+CD4+、CD3+CD8+ and so on) in peripheral blood by cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ou-Yang, M.D., Principal Investigator — The First Affiliated Hospital, Guangzhou Medical University，China
Locations (1):
- The First Affiliated Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen L, He Z, Qin L, Li Q, Shi X, Zhao S, Chen L, Zhong N, Chen X. Antitumor effect of malaria parasite infection in a murine Lewis lung cancer model through induction of innate and adaptive immunity. PLoS One. 2011;6(9):e24407. doi: 10.1371/journal.pone.0024407. Epub 2011 Sep 9. PMID 21931708